CLINICAL TRIAL: NCT07179991
Title: Desmopressin Effect on Platelet Function Assessment by Thromboelastography (TEG 6) in Cardiac Surgery
Brief Title: DDAVP Effect by TEG6 in Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Satoru Fujii, Anesthesiologist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: DDAVP TEG6
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Intraoperative Bleeding
Keywords: Desmopressin; Cardiopulmonary bypass
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Desmopressin after protamine reversal: Desmopressin will be given to participants at a dose of 0.3mcg/kg after protamine reversal at the end of cardiopulmonary bypass (CPB).
  Interventions: Drug: Desmopressin after protamine reversal

INTERVENTIONS:
Drug: Desmopressin after protamine reversal — Desmopressin will be given to participants at a dose of 0.3mcg/kg after protamine reversal at the end of cardiopulmonary bypass (CPB).
  Platelet function will be assessed by TEG (Thromboelastography) platelet mapping at the following points:
  1. T1 TEG6s: after arterial line insertion before skin incision.
  2. T2 TEG6s: after protamine (baseline function after CPB)
  3. T3 TEG6s: 30 minutes after desmopressin
  4. T4 TEG6s: 6 hours after (intensive care unit) ICU admission
  5. T5 TEG6s: 24hours after ICU admission

SUMMARY:
Cardiopulmonary bypass (CPB) is a process that uses a pump that temporarily takes over the function of the heart and lungs during cardiac surgery to maintain blood circulation and oxygenation. Using CPB during cardiac surgery can result in complications with blood clotting. Blood clotting is achieved when molecules in the blood, called platelets, are able to form together with the help of other clotting factors to form a clot. A drug called desmopressin (DDAVP) is used to help blood clot properly by increasing the amount of clotting factors in the blood. Several studies have shown that desmopressin has the ability to reduce the amount of blood transfusions needed for cardiac surgery patients in the postoperative period. At LHSC desmopressin is frequently requested by Cardiac Surgeons and Anesthesiologists to stop bleeding and promote blood clotting where required. A test called TEG6s platelet mapping is a blood test used to help manage the use of blood products by being able to provide information on platelet function and blood clotting activity. At the moment, there is a lack of information regarding the use of TEG6s platelet mapping to analyze the effect of desmopressin on blood clotting in cardiac surgery patients after CPB. The purpose of this study is to investigate the dose-related effects of desmopressin on platelet function in patients undergoing cardiac surgery with CPB. By using TEG6s platelet mapping, this study aims to observe dynamic changes in platelet function following desmopressin administration at various time points in the perioperative and postoperative periods.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) during cardiac surgery is frequently complicated by disturbances in coagulation parameters and platelet function. Desmopressin (DDAVP) has been utilized to enhance platelet adhesion and aggregation by increasing plasma levels of von Willebrand factor (vWF) and factor VIII that plays a crucial role in blood clotting. Several studies demonstrated a positive effect of DDAVP in hemostasis (particularly in patients with qualitative platelet dysfunction), reduced blood transfusion and bleeding in the post operative period.

Viscoelastic testing, specifically TEG (Thromboelastography) platelet mapping and TEG6s and have been shown to be helpful in managing the use of blood products, fresh frozen plasma (FFP), platelets and fibrinogen, in coagulopathic patient post cardiopulmonary bypass. Desmopressin is given at a dose 0.3 micrograms/kg intravenously over 15 to 30 minutes as a standard dose in cardiac surgery, up to 20 mcg which is the United States Food and Drug Administration (US FDA) recommended dose for Hemophilia treatment and the most commonly cited dose used in cardiac surgery after cardiopulmonary bypass. The TEG6s platelet mapping shows baseline platelet function and receptor-specific platelet function and inhibition. This assessment is based on four different assays including Koalin, Activator F, ADP (Adenosine Diphosphate), AA (Arachidonic Acid). At the current time there is limited literature looking at the qualitative effect of desmopressin on platelet function using TEG6s platelet mapping analysis. The purpose of this study is to investigate the dose-related effects of desmopressin on platelet function in patients undergoing cardiac surgery. By using TEG6s platelet mapping we aim to observe dynamic changes in platelet function following desmopressin administration at various time points in perioperative and postoperative periods.

Informed, written consent will be obtained prior to the start of surgery.

Participants that are enrolled in this study will have their surgery proceed according to plan and will be placed under general anesthesia using standard of care practices. Cardiopulmonary bypass will be implemented in accordance with standard of care practices. Desmopressin will be given to participants at a dose of 0.3mcg/kg, up to 20 mcg after protamine reversal at the end of cardiopulmonary bypass.

Platelet function will be assessed by TEG platelet mapping at the following points:

1. T1 TEG6s: after arterial line insertion before skin incision.
2. T2 TEG6s: after protamine (baseline function after CPB)
3. T3 TEG6s: 30 minutes after desmopressin
4. T4 TEG6s: 6 hours after (intensive care unit) ICU admission
5. T5 TEG6s: 24hours after ICU admission

This will involve drawing 4 ml of blood from patients at each of the above time points (5 blood draws total), in a dark green-top (Sodium Heparin) Vacutainer® tube by the Cardiac Anesthesiologist who will be also running the test on the TEG Machine. The study team will also collect information such as participant age, biological sex, height, weight, medications, medical history, surgical details, results of preoperative and postoperative blood work, and details of their postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Undergoing elective cardiac surgery with cardiopulmonary bypass
3. Able to provide informed consent

Exclusion Criteria:

1. Hyponatremia
2. Allergy to desmopressin or its components
3. History of coronary artery disease with thrombosis
4. Recent history of thromboembolic events (Stroke/TIA/DVTs)
5. Severe Renal Impairment Creatinine Clearance<30 ml/min
6. Inability to communicate in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational, single centre study being conducted at London Health Sciences Centre (LHSC) with adults undergoing elective cardiac surgery with cardiopulmonary bypass to investigate the dose-related effects of desmopressin on platelet function in patients undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in platelet function due to desmopressin administration after cardiopulmonary bypass | After arterial line insertion - 24 hours after admission to the intensive care unit
  This will be measured by TEG6s platelet mapping.

SECONDARY OUTCOMES:
Impact of desmopressin on transfusion products required | After arterial line insertion - 24 hours after admission to the intensive care unit
  This will be measured by recording the amount of blood products required for transfusion.
Impact of desmopressin on chest drainage | After arterial line insertion - 24 hours after admission to the intensive care unit
  This will be measured by recording the fluid drained from the chest of participants

CONTACTS AND LOCATIONS:
Overall Officials: Satoru Fujii, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mongan PD, Hosking MP. The role of desmopressin acetate in patients undergoing coronary artery bypass surgery. A controlled clinical trial with thromboelastographic risk stratification. Anesthesiology. 1992 Jul;77(1):38-46. doi: 10.1097/00000542-199207000-00007. PMID 1610009
- [Background] Ozkisacik E, Islamoglu F, Posacioglu H, Yagdi T, Basarir S, Omay SB, Ozbaran M, Buket S. Desmopressin usage in elective cardiac surgery. J Cardiovasc Surg (Torino). 2001 Dec;42(6):741-7. PMID 11698939
- [Background] Jahangirifard A, Mirtajani SB, Madadi F. Effect of Desmopressin on Bleeding After Heart Surgeries: A Narrative Review. Anesth Pain Med. 2023 Mar 10;13(2):e133894. doi: 10.5812/aapm-133894. eCollection 2023 Apr. PMID 37645010
- [Background] Wademan BH, Galvin SD. Desmopressin for reducing postoperative blood loss and transfusion requirements following cardiac surgery in adults. Interact Cardiovasc Thorac Surg. 2014 Mar;18(3):360-70. doi: 10.1093/icvts/ivt491. Epub 2013 Nov 21. PMID 24263581
- [Background] Despotis GJ, Levine V, Saleem R, Spitznagel E, Joist JH. Use of point-of-care test in identification of patients who can benefit from desmopressin during cardiac surgery: a randomised controlled trial. Lancet. 1999 Jul 10;354(9173):106-10. doi: 10.1016/S0140-6736(98)12494-7. PMID 10408485
- [Background] Agarwal S, Abdelmotieleb M. Viscoelastic testing in cardiac surgery. Transfusion. 2020 Oct;60 Suppl 6:S52-S60. doi: 10.1111/trf.16075. Epub 2020 Sep 21. PMID 32955756
- [Background] Meco M, Montisci A, Giustiniano E, Greco M, Pappalardo F, Mammana L, Panisi P, Roscitano C, Cirri S, Donatelli F, Albano G. Viscoelastic Blood Tests Use in Adult Cardiac Surgery: Meta-Analysis, Meta-Regression, and Trial Sequential Analysis. J Cardiothorac Vasc Anesth. 2020 Jan;34(1):119-127. doi: 10.1053/j.jvca.2019.06.030. Epub 2019 Jun 28. PMID 31445833
- [Background] Li C, Zhao Q, Yang K, Jiang L, Yu J. Thromboelastography or rotational thromboelastometry for bleeding management in adults undergoing cardiac surgery: a systematic review with meta-analysis and trial sequential analysis. J Thorac Dis. 2019 Apr;11(4):1170-1181. doi: 10.21037/jtd.2019.04.39. PMID 31179059
- [Background] Jin L, Ji HW. Effect of desmopressin on platelet aggregation and blood loss in patients undergoing valvular heart surgery. Chin Med J (Engl). 2015 Mar 5;128(5):644-7. doi: 10.4103/0366-6999.151663. PMID 25698197
- [Background] Salmenpera M, Kuitunen A, Hynynen M, Heinonen J. Hemodynamic responses to desmopressin acetate after CABG: a double-blind trial. J Cardiothorac Vasc Anesth. 1991 Apr;5(2):146-9. doi: 10.1016/1053-0770(91)90328-q. PMID 1863726
- [Background] Cattaneo M, Harris AS, Stromberg U, Mannucci PM. The effect of desmopressin on reducing blood loss in cardiac surgery--a meta-analysis of double-blind, placebo-controlled trials. Thromb Haemost. 1995 Oct;74(4):1064-70. PMID 8560415
- [Background] Desborough MJ, Oakland K, Brierley C, Bennett S, Doree C, Trivella M, Hopewell S, Stanworth SJ, Estcourt LJ. Desmopressin use for minimising perioperative blood transfusion. Cochrane Database Syst Rev. 2017 Jul 10;7(7):CD001884. doi: 10.1002/14651858.CD001884.pub3. PMID 28691229
- [Background] Rogers AL, Allman RD, Fang X, Kindell LC, Nifong LW, Degner BC, Akhter SA. Thromboelastography-Platelet Mapping Allows Safe and Earlier Urgent Coronary Artery Bypass Grafting. Ann Thorac Surg. 2022 Apr;113(4):1119-1125. doi: 10.1016/j.athoracsur.2021.07.068. Epub 2021 Aug 24. PMID 34437860
- [Background] Sivapalan P, Back AC, Ostrowski SR, Ravn HB, Johansson PI. Transfusion requirements in elective cardiopulmonary bypass surgery patients: predictive value of Multiplate and Thromboelastography (TEG) Platelet Mapping Assay. Scand J Clin Lab Invest. 2017 Sep;77(5):345-351. doi: 10.1080/00365513.2017.1325000. Epub 2017 May 24. PMID 28537454
- [Background] Agarwal S, Johnson RI, Kirmani BH. Pre- and Post-Bypass Platelet Function Testing With Multiple Electrode Aggregometry and TEG Platelet Mapping in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2015 Oct;29(5):1272-6. doi: 10.1053/j.jvca.2015.01.028. Epub 2015 Jan 16. PMID 25987196